CLINICAL TRIAL: NCT07316114
Title: A Prospective Observational Study of Patients Receiving Dupilumab for Chronic Spontaneous Urticaria
Brief Title: A Study to Describe the Real-world Effectiveness, Safety and Patterns of Use of Dupilumab in Patients With Chronic Spontaneous Urticaria
Acronym: DEDICATION
Status: Not yet recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18182; U1111-1331-3693 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-12-08; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dupilumab — This study will not administer any treatment, only observe the treatment as prescribed in real world clinical practice.

SUMMARY:
This is a decentralized study designed to describe the real-world effectiveness, safety, and patterns of use of dupilumab in patients with chronic spontaneous urticaria (CSU). This study will be conducted in the United States and will collect data available from participants' medical files, other items routinely collected during disease management in clinical practice, and patient-reported outcomes related to disease, work productivity, quality of life, and CSU-related hospitalizations.

Participation in this study is the patient's own choice and is entirely voluntary. The treating physician prescribes dupilumab treatment as part of routine care, independently of the study. Once the decision to prescribe dupilumab is made by the treating physician, patients can self-screen and will be contacted by the Virtual Research Coordination Center to determine potential study eligibility. Patients will be enrolled if they provide an informed consent and meet all inclusion criteria and none of the exclusion criteria.

The duration of the study for each participant is 24 months. All patients will be followed for 24 months or until death, loss to follow-up, or withdrawal, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years or older at the time of informed consent/assent.
* Physician decision to treat the patient with dupilumab for chronic spontaneous urticaria (CSU) made prior to and independently of the patient's participation in the study.
* Patient is able to understand and complete study-related questionnaires.
* Patients and/or parent/legally authorized representative provide voluntary informed consent and/or assent to participate in the study before inclusion in the study.

Exclusion Criteria:

* Patients who have a contraindication to dupilumab according to the approved prescribing information label.
* Any condition that the treating physician or virtual Investigator believes may interfere with the patient's ability to participate in the study, such as short life expectancy, substance abuse, severe cognitive impairment, or other comorbidities that can predictably prevent the patient from completing the schedule of assessments.
* Patients currently participating in any interventional clinical trial.
* Prior use of dupilumab within 6 months of the baseline assessment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study aims to enroll approximately 10% to 20% adolescents (that is, participants aged 12 to 17 years) of the total 400 participants. If the adolescent enrollment target is not met toward the end of the period, adult enrollment may be temporarily paused to allow more adolescents to enroll.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-11-24 (Estimated); Study Completion 2029-11-22 (Estimated)

PRIMARY OUTCOMES:
Summary of Sociodemographic Characteristics | Baseline
  Sociodemographic and clinical characteristics, including but not limited to month and year of birth, age, sex, race, ethnicity, IgE levels, employment status, height, weight, and smoking status will be collected.
Summary of Medical History of Chronic Spontaneous Urticaria (CSU) | Baseline
  Medical history of CSU, including but not limited to CSU status and CSU treatment history will be collected.
Summary of Type of Baseline Comorbidities | Baseline
  Type of baseline comorbidities including atopic and non-atopic will be collected.
Summary of Type of Concomitant Medication | Baseline
  Type of concomitant medication will be collected.
Summary of Healthcare Provider Specialties | Baseline
  Healthcare practitioner's information (related to CSU treatment) and specialty (example, dermatology physician, dermatology nurse practitioner, dermatology physician assistant, allergy/immunology physician, allergy/immunology nurse practitioner, allergy/immunology physician assistant) will be collected.
Summary of Dupilumab Dosing Regimen | Baseline
  Summary of dupilumab dosing regimen, duration of treatment, time to discontinuation and other discontinuation details, and treatment modifications/interruptions and reasons will be collected.
Summary of Treatments Used After Discontinuation | Baseline
  Summary of treatments used after discontinuation will be collected.
Summary of Participants Re-treated with Dupilumab and Reason | Baseline
  Summary of participants re-treated with dupilumab and reason will be collected.

SECONDARY OUTCOMES:
Change from Baseline in Disease Activity | Baseline to up to 24 months
  Change from baseline in disease activity as assessed by Urticaria Activity Score over 7 days (UAS7) and Urticaria Control Test (UCT) scores.
Dupilumab Treatment Details: Summary of Participants who Achieve Response Thresholds | Baseline to up to 24 months
  Summary of participants who achieve response thresholds, including onset of response, peak response, recapture response will be collected to evaluate the real-world long-term effectiveness of dupilumab for the treatment of CSU.
Dupilumab Treatment Details: Summary of Participants who Achieve Disease Control Thresholds | Baseline to up to 24 months
  Summary of participants who achieve disease control thresholds will be collected to evaluate the real-world long-term effectiveness of dupilumab for the treatment of CSU.
Dupilumab Treatment Details: Durability of Response During and After Discontinuation of Dupilumab | Baseline to up to 24 months
  Durability of response will be assessed by using Urticaria Activity Score over 7 days (UAS7). It is based on scoring wheals (hive severity score) and itch (itch severity score) separately on a scale of 0 (no signs/symptoms) to 3 (intense signs/symptoms) over 7 days. The final score is calculated by adding together the daily scores, which can range from 0 to 6, for 7 days. This results in a maximum total score of 42, and a minimum possible score of 0.
Dupilumab Treatment Details: Duration of Disease Control | Baseline to up to 24 months
  Duration of disease control prior to and after discontinuation of dupilumab will be assessed.
Change from Baseline in Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL) for Adult Participants | Baseline to up to 24 months
  The CU-Q2oL is a patient-reported outcome measure designed to assess the impact of chronic urticaria on various aspects of a patient's life. It includes questions that evaluate physical symptoms, emotional well-being, daily activities, sleep quality, and treatment satisfaction. Responses are scored on a 5-point Likert scale, reflecting the overall QoL impairment, with higher scores indicating greater negative impact.
Change from Baseline in Dermatology Life Quality Index (DLQI) for Participants 16 years of Age or Older | Baseline to up to 24 months
  The DLQI is a 10-question, patient-reported outcome measure designed to assess the impact of skin diseases on the QoL.24 It covers domains such as symptoms, emotional well-being, leisure activities, school performance, personal relationships, and treatment burden. Each question is scored from 0 to 3, with a total score ranging from 0 to 30, where higher scores indicate greater impairment.
Change from Baseline in Children's Dermatology Life Quality Index (CDLQI) for Participants 15 Years of Age or Younger | Baseline to up to 24 months
  The CDLQI is a 10-question, patient-reported outcome measure designed to assess the impact of skin diseases on the QoL.24 It covers domains such as symptoms, emotional well-being, leisure activities, school performance, personal relationships, , and treatment burden. Each question is scored from 0 to 3, with a total score ranging from 0 to 30, where higher scores indicate greater impairment.
Change from Baseline in Work Productivity and Activity Impairment: Chronic urticaria (WPAI:CU) for Adult Participants | Baseline to up to 24 months
  The WPAI:CU is a 6-item PRO instrument that measures the effect of a condition on productivity during work and regular activities in the 7 days prior to completion. The instrument comprises 4 domains: absenteeism, presenteeism, overall work impairment, and activity impairment due to chronic urticaria. WPAI:CU outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change from Baseline in Treatment satisfaction (TSQM-9) for Adult Participants | Baseline to up to 24 months
  The TSQM-9 is a 9-item PRO measure designed to evaluate satisfaction with medication across 3 domains: effectiveness, side effects, and convenience.27 It uses a 5- or 7-point Likert scale to score responses, which are then transformed to a 0-100 scale, with higher scores indicating greater satisfaction.
CSU-related Hospitalization | Baseline to up to 24 months
  CSU-related hospitalization including number of hospital visits, number of emergency department visits, number of specialist visits will be collected.
Number of Particiapants Experiencing Adverse Events | Baseline to up to 24 months
  Number of participants experiencing AEs will be assessed.
Number of Participants Experiencing Serious Adverse Events (SAEs) | Baseline to up to 24 months
  Number of participants experiencing SAEs will be assessed.
Number of Participants Experiencing Adverse Events of Special Interest (AESI) | Baseline to up to 24 months
  Number of participants experiencing AESI will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual Research Coordination Center, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org